CLINICAL TRIAL: NCT05826847
Title: Effect of Prone Positioning and Abdominal Binding on Lung and Muscle Protection in ARDS Patients With ICU-acquired Weakness Transitioning From Controlled to Spontaneous Breathing
Brief Title: Prone Positioning and Abdominal Binding on Lung and Muscle Protection in ARDS Patients During Spontaneous Breathing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Rodrigo Cornejo, Full Professor, University of Chile
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1221829
Record Dates: First submitted 2023-03-06; First posted 2023-04-24 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation Complication; ICU Acquired Weakness
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Three phase-study:
  1. Multimodal physiological description
  2. Randomized crossover trial
  3. Pilot randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Sham Comparator): ARDS patients at spontaneous breathing onset on pressure support ventilation mode in supine position at 45º degrees, performed under standard PEEP according to ARDSNet strategy and individualized PEEP applied in random order.
  Interventions: Procedure: Control
- Prone Positioning (Experimental): ARDS patients at spontaneous breathing onset on pressure support ventilation mode in prone position, performed under standard PEEP according to ARDSNet strategy and individualized PEEP applied in random order.
  Interventions: Procedure: Prone Positioning
- Thoracoabdominal Binding (Experimental): ARDS patients at spontaneous breathing onset on pressure support ventilation mode in supine position at 45º degrees using thoracoabdominal binding with the binder's upper edge above the costal margin, performed under standard PEEP according to ARDSNet strategy and individualized PEEP applied in random order.
  Interventions: Procedure: Thoracoabdominal Binding

INTERVENTIONS:
Procedure: Prone Positioning — Prone positioning will be performed according to ICU local protocol with trained provider teams.
  Arms: Prone Positioning
Procedure: Thoracoabdominal Binding — Thoracoabdominal binding will be used in semi-recumbent position (supine at 45º) and titrated to obtain a 20-30% decrease in chest wall compliance and 1-3 cm H2O increase in end-expiratory gastric pressure during steady-state breathing
  Arms: Thoracoabdominal Binding
Procedure: Control — ARDS patients at spontaneous breathing onset on pressure support ventilation mode in supine position at 45º degrees, performed under standard PEEP according to ARDSNet strategy and individualized PEEP applied in random order.
  Arms: Control Group

SUMMARY:
Ventilator-induced diaphragmatic dysfunction and intensive care unit (ICU)-acquired weakness are two consequences of prolonged mechanical ventilation and critical illness in patients with acute respiratory distress syndrome (ARDS). Both complicate the process of withdrawing mechanical ventilation, increase hospital mortality and cause chronic disability in survivors. During transition from controlled to spontaneous breathing, these complications of critical illness favor an abnormal respiratory pattern and recruit accessory respiratory muscles which may promote additional lung and muscle injury. The type of ventilatory support and positioning may affect the muscle dysfunction and patient-self-inflicted lung injury at spontaneous breathing onset. In that regard, ARDS patients with ventilator-induced diaphragmatic dysfunction and ICU-acquired weakness who are transitioning from controlled to partial ventilatory support probably present an abnormal respiratory pattern which exacerbates lung and muscle injury. Physiological-oriented ventilatory approaches based on prone positioning or semi recumbent positioning with abdominal binding at spontaneous breathing onset, could decrease lung and muscle injury by favoring a better neuromuscular efficiency, and preventing intense inspiratory efforts and high transpulmonary driving pressures, as well as high-magnitude pendelluft. In the current project, in addition to perform a multimodal description of the severity of ventilator-induced diaphragmatic dysfunction and ICU-acquired weakness in prolonged mechanically ventilated ARDS patients, prone positioning and supine plus thoracoabdominal binding at spontaneous breathing onset will be evaluated.

DETAILED DESCRIPTION:
Study protocol will have three steps. The first step is a multimodal description to characterize ICU acquired weakness and ventilator-induced diaphragm dysfunction in prolonged mechanically ventilated ARDS patients at spontaneous breathing onset. The second step is a crossover clinical trial to test different ventilatory approaches oriented to improve physiological variables related to lung injury and diaphragm performance. The third step is a randomized controlled trial to test the effect of the previous ventilatory approaches on lung inflammatory response and biomarkers of lung and muscular injury.

FIRST STEP: A multimodal physiological description will be performed in pressure support ventilation mode at spontaneous breathing onset. The assessments will include conventional electromyography; electrical activity of the diaphragm; ultrasound of respiratory and non-respiratory muscles; respiratory flow; tidal volume; airway, esophageal and gastric pressures; and hemodynamic and electric impedance tomography monitoring at the end of 2-hours of spontaneous breathing period.

SECOND STEP: A controlled randomized crossover trial will assign patients to three strategies of 2-hours period on pressure support ventilation mode: A.- Control group: supine at 45º, B.- Thoracoabdominal binding: supine at 45º plus thoracoabdominal binding, C.- Prone positioning (without thoracoabdominal binding). These strategies will be performed under standard positive end-expiratory pressure (PEEP) (ARDSNet strategy) and individualized PEEP (obtained at the lowest combination of collapse and overdistension according to electrical impedance tomography), applied in random order. Therefore, each patient will receive the six approaches, with washout periods of 15-minutes in assisted/controlled ventilation.

THIRD STEP: Patients will be randomized to one of the three ventilatory strategies previously defined, A.- Control group: supine at 45º, B.- Thoracoabdominal binding: supine at 45º plus abdominal binding, C.- Prone positioning. These three strategies will be applied under standard PEEP (ARDSNet strategy). Between crossover and pilot randomized controlled trial, the patients will remain under moderate sedation in pressure support ventilation mode receiving an individualized PEEP level.

ELIGIBILITY:
Inclusion Criteria:

* Adult ARDS patients with moderate-severe ARDS on controlled protective mechanical ventilation for more than 3 days
* Stable hemodynamics
* Level of consciousness enough to initiate spontaneous breathing

Exclusion Criteria:

* Unstable hemodynamics
* Tracheostomy
* Abnormal level of consciousness
* Central nervous system injury
* Esophageal varices
* Pregnancy
* Contraindications for installation of electrical impedance tomography or ultrasound assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
(Second Phase) High-Magnitude Pendelluft | Two hours on each ventilatory strategy during phase 2
  Frequency of high-magnitude pendelluft monitored by electrical impedance tomography
(Third Phase) Change in Inflammatory Biomarkers Measured by ELISA (IL-6, IL-8, TNF-α, IFN-γ, IL-18, IL-1β, Caspase-1, RAGE, Angiopoietin-1 and 2) and change in oxidative stress related biomarkers (F2 isoprostane) | At baseline and after 24 hours of each ventilatory strategy during phase 3
  ELISA-based detection of inflammatory biomarkers (absolute and ratios) and oxidative stress related biomarkers (absolute and ratios) measured in plasma and in exhaled breath condensate
(Third Phase) Change in Regional Lung Inflammation | At baseline and after 24 hours of each ventilatory strategy during phase 3
  Regional lung inflammation will be evaluated with dynamic positron emission tomography/computed tomography of fluoro-2-deoxy-D-glucose (18F-FDG) net uptake rate
(Third Phase) Change in Fast-Twitch Skeletal Muscle Troponin I Measured by ELISA | At baseline and after 24 hours of each ventilatory strategy during phase 3
  ELISA-based detection of fast-twitch skeletal muscle troponin I measured in plasma

SECONDARY OUTCOMES:
(Second Phase) Respiratory Mechanics Variables | Two hours on each ventilatory strategy during phase 2
  Esophageal pressure swing, transdiaphragmatic pressure and transpulmonary driving pressure measured by a esophageal/gastric catheter
(Third Phase) Change in High-Magnitude Pendelluft | At baseline and after 24 hours of each ventilatory strategy during phase 3
  Frequency of high-magnitude pendelluft monitored by electrical impedance tomography
(Third Phase) Change in Respiratory Mechanics Variables | At baseline and after 24 hours of each ventilatory strategy during phase 3
  Esophageal pressure swing, transdiaphragmatic pressure and transpulmonary driving pressure measured by a esophageal/gastric catheter
(Third Phase) Change in Neuromechanical Coupling of Diaphragm | At baseline and after 24 hours of each ventilatory strategy during phase 3
  Change in neuromechanical coupling of diaphragm, which corresponds to the ratio between transdiaphragmatic pressure and electrical activity of the diaphragm measured by a esophageal/gastric catheter

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Cornejo, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Independencia, Chile

IPD SHARING:
Plan to Share IPD: No